CLINICAL TRIAL: NCT05209126
Title: Impact of an Acute Beetroot Ingestion on Neuromuscular Performance in Female Rugby Players
Brief Title: Impact of Beetroot Juice Ingestion on Female Rugby Performance
Acronym: BEETJUICERUGBY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: University of Seville (Other); Universidad Complutense de Madrid (Other); University of Alcala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Universidad_FranciscoVitoria
Record Dates: First submitted 2022-01-14; First posted 2022-01-26 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-01

CONDITIONS: Nitric Oxide; Placebo
Keywords: dietary supplements; nitrate; sports performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot supplementation (Experimental): One serving 140 mL of beetroot juice (12.8 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 3 h before initiating the testing session.
  Interventions: Dietary Supplement: Beetroot juice
- Placebo supplementation (Placebo Comparator): One serving 140 mL of beetroot juice placebo (0.08 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 3 h before initiating the testing session.
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Acute effects of beetroot juice ingestion on neuromuscular performance in female rugby players
  Other Names: Nitrate precursors

SUMMARY:
Rugby is a team sport characterized by high-intermittent efforts, due to the importance of realizing intermittent and explosive efforts in rugby the use of nutritional strategies such as beetroot ingestion should be explored with the aim to enhance the capacity for repeating high-intensity actions in female players.

DETAILED DESCRIPTION:
Rugby is a team sport characterized by high-intermittent efforts, thus, to the importance of realizing intermittent and explosive efforts in field hockey is crucial. For this reason, the use of nutritional strategies in field hockey should be explored with the aim to enhance the capacity for repeating high-intensity actions. However, scientific evidence supports only a few numbers of dietary supplements that have reported good evidence for improving sports performance, between we can mention beetroot juice supplementation with doses > 5 mmol of NO3-. Beetroot juice is a NO3- precursor with recognized effectiveness to elicit performance due to different physiological mechanisms associated with its ingestion such as increment in vasodilatation, skeletal muscle contractility, or delaying fatigue development that could be linked with an enhance or performance in team-sports athletes. However, the majority of the studies has been realized in male athletes being female athletes underrepresented in beetroot juice supplementation research. Thus, the aim of this study was to analyze the effects of beetroot juice ingestion on neuromuscular performance in female rugby players.

ELIGIBILITY:
Inclusion Criteria:

* More than 5 years of rugby training experience.
* Active rugby player

Exclusion Criteria:

* Concurrently participating in other studies.
* Contraindications to beetroot juice ingestion.
* Physical limitations, health problems, or musculoskeletal injuries.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study analyze the effects of beetroot juice ingestion in female rugby players.
Enrollment: 13 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in Bronco Aerobic Fitness Test | 1-week
  Time to complete test using photocell timing gates

SECONDARY OUTCOMES:
Changes in maximal isometric handgrip strength (kg) | 1-week
  Using a hand-held dynamometer
Changes in maximal jump height (cm) | 1 week
  Maximal jump height using a contact platform
Changes in 30-meters sprint time (s) | 1 week
  Time to complete 30-m sprints using photocell timing gates
Changes in rate of perceived exertion scale | 1-week
  Differences between placebo and beetroot juice in rate of perception exertion scale
Changes in side effects questionnarie | 1-week
  Differences between placebo and beetroot juice in side effects health aspects

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid
  - Universidad Francisco de Vitoria, Madrid